CLINICAL TRIAL: NCT04293133
Title: Final Height in Patients With Congenital Adrenal Hyperplasia
Brief Title: Final Height in Patients With CAH
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Mohammed Kamel El-Desouky Ashour, Final height in patients with congenital adrenal hyperplasia, Ain Shams University
Other Study IDs: CAH
Record Dates: First submitted 2020-03-02; First posted 2020-03-03 (Actual); Last update posted 2020-03-03 (Actual); Status verified 2020-03

CONDITIONS: Congenital Adrenal Hyperplasia
MeSH Terms: conditions — Adrenal Hyperplasia, Congenital

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Congenital adrenal hyperplasia (CAH) is the most common inherited disorder in the adrenal gland in children. Growth is usually affected in CAH patients either due to the disease itself or treatment consequences.

DETAILED DESCRIPTION:
CAH comprises a group of autosomal recessive disorders caused by a deficiency of one of five enzymes needed for the synthesis of cortisol leading to defect in cortisol synthesis with or without aldosterone deficiency and an increase in the production of adrenocorticotropic hormone through negative feedback.

The most common form is 21-hydroxylase deficiency (21OHD), which forms more than 90 % of the cases.

In classic CAH, 75% of the patients have the salt wasting (SW) and 25% have the non salt-wasting phenotype (NSW).There are no clinical signs at birth in male infants and in female patients, CAH is suspected shortly after birth if there is genital ambiguity, ranging from slight clitromegaly to complete masculinization with acceleration of growth and pubertal development.

The non-classic (late onset) form of CAH is a less severe form of 21OHD, and is diagnosed later in life.

Final height in early and late onset patients has been reported as diminished (Hauffa et al, 1997).This could be attributed to androgen excess or treatment with steroids. Androgen excess can occur at any age leading to accelerated growth, early epiphyseal closure and compromised final adult height.

Despite that all forms of CAH differ in their degree of enzymatic deficiency, they all represent a therapeutic challenge to pediatric endocrinologists attempting to optimize growth.

ELIGIBILITY:
Inclusion Criteria:

* Patients having a documented history of classical CAH.

Exclusion Criteria:

* Patients with non classical CAH.
* Patients treated with growth hormone.
* Chronic use of medications unrelated to CAH which may affect growth like immunosuppressive drugs like azathioprine and drugs that affect growth hormone release like octreotide, pegvisomant, bromocriptine and cabergoline.
* Other chronic diseases that may affect growth like heart disease, inflammatory bowel disease and renal disease.
* Other causes of adrenal insufficiency.

Max Age: 18 Years | Sex: All
Age Groups: Child, Adult
Study Population: Patients having a documented history of classical CAH.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2020-03-11 (Estimated); Primary Completion 2020-08-11 (Estimated); Study Completion 2020-09-11 (Estimated)

PRIMARY OUTCOMES:
Final height in patients with congenital adrenal hyperplasia | Baseline
  Target height(TH) will be calculated using the formula: [maternal height + paternal height - 13 cm for girls and + 13 cm for boys]/2

CONTACTS AND LOCATIONS:
Overall Officials: Rana Ahmed, Principal Investigator — Ain Shams University

REFERENCES:
- [Background] Cole TJ, Freeman JV, Preece MA. Body mass index reference curves for the UK, 1990. Arch Dis Child. 1995 Jul;73(1):25-9. doi: 10.1136/adc.73.1.25. PMID 7639544
- [Background] Charmandari E, Brook CG, Hindmarsh PC. Classic congenital adrenal hyperplasia and puberty. Eur J Endocrinol. 2004 Nov;151 Suppl 3:U77-82. doi: 10.1530/eje.0.151u077. PMID 15554890